CLINICAL TRIAL: NCT01452737
Title: 2L Golytely and Oral Bisacodyl 15 mg Versus 4L Golytely Regimen for Inpatient Colonoscopy Bowel Preparation: A Randomized, Non-Inferiority Open Trial
Brief Title: Comparing 4L Golytely to 2L Golytely With 15mg Bisacodyl Regimens for Inpatient Colonic Preparation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H11-02318
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Colonoscopy
Keywords: colonoscopy; bowel preparation; Golytely
MeSH Terms: interventions — Golytely; Bisacodyl

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 2L Golytely/15mg bisacodyl (Experimental): Subjects will be asked to take 2L Golytely + 15mg bisacodyl for bowel prep the day before colonoscopy.
  Interventions: Drug: 2L Golytely/bisacodyl
- Standard bowel prep (Active Comparator): Subject will receive standard bowel prep (4L Golytely) prior to colonoscopy.
  Interventions: Drug: Standard Bowel Prep

INTERVENTIONS:
Drug: Standard Bowel Prep — Subjects will be asked to take 4L of Golytely the day prior to procedure.
  Arms: Standard bowel prep
Drug: 2L Golytely/bisacodyl — Subjects will be asked to take 2L Golytely and 15mg bisacodyl the day prior to procedure.
  Arms: 2L Golytely/15mg bisacodyl

SUMMARY:
The investigators wish to compare the efficacy and patient tolerability of a preparation consisting of 2L Golytely (PEG + electrolytes) plus 15mg of bisacodyl vs the standard preparation of 4L Golytely. The investigators hypothesize that 2L Golytely with 15mg bisacodyl will show similar bowel cleansing efficacy while offering better tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients undergoing colonoscopy
* Age 19 or over

Exclusion Criteria:

* Unable to provide informed consent
* Patients with constipation
* Patients with suspected bowel obstruction or severe inflammatory bowel disease
* Same-day colonoscopy
* Intensive/critical care patient
* History of colorectal resection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Difference in Boston Bowel Preparation Scale & Ottawa Bowel Preparation Scale between the two groups | 30min
  These are established rating scales to evaluate the quality of bowel prep. The ratings will be compared between the two groups.

SECONDARY OUTCOMES:
Difference in the number of participants who develop distress symptoms from bowel prep (and the type) between the two groups | 20hours
  Number of participants who develop distress symptoms from bowel prep, and the type of distress symptoms will be compared between the two groups
Difference in the absolute number/percentage of participants in the two groups who find the bowel prep experience easy, acceptable, difficult, very difficult, or unable to complete. | 20hours
  Participants will be asked to rate their bowel prep experience (based on ease of use) on a Likert scale. The number of participants in each level will subsequently be quantified (n, %) and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Enns, Dr., Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada